CLINICAL TRIAL: NCT01097473
Title: Effects of Long Term Physical Training Once a Week on Fitness and Quality of Life in Elderly Asthmatics
Brief Title: Long Term Physical Training in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Andreas Meyer, Krankenhaus St. Kamillus, Mönchengladbach, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AM-001
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2010-04-01 (Estimated); Status verified 2010-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise training (Active Comparator): Subjects participate in a once weekly supervised exercise training group, duration of 60 min.
  Interventions: Procedure: Exercise training
- Control (No Intervention): Control group receives no intervention

INTERVENTIONS:
Procedure: Exercise training — Exercise training in outpatient sport groups once weekly with a duration of 60 min each
  Arms: Exercise training

SUMMARY:
This controlled study is undertaken to investigate the effects of a long term outpatient training program on physical fitness and quality of life in elderly asthmatics.

DETAILED DESCRIPTION:
Physical training is well known to support a healthy lifestyle. Patients with asthma are often unnecessarily restricted of physical activities or avoid exercise due to the unpleasant experience of exercise-induced dyspnea. As a consequence both children and adults with asthma are less fit than their peers. Like in healthy individuals, regular training supports health in asthmatics. In short-term training programs improvements of physical capabilities have been achieved in children and young adults with asthma. Programs of longer durations than 3 months have not been published in controlled trials. Effects of exercise training on quality of life in adult asthmatics are lacking.

ELIGIBILITY:
Inclusion Criteria:

* physician diagnosed asthma
* non-smoker
* stable condition
* informed consent

Exclusion Criteria:

* participation in pulmonary rehabilitation in the past 12 months prior to study inclusion
* unability to attend training sessions on a regular basis for one year
* symptomatic coronary heart disease
* uncontrolled heart failure
* hemodynamically relevant cardiac rhythm disorders
* hemodynamically relevant cardiac valvular disorders
* uncontrolled arterial hypertension
* hypercapnic respiratory failure
* severe hypoxemia (i.e. PaO2 <50 mm Hg resp. SaO2 <80% at rest)
* history of decompensated right heart failure
* pulmonary arterial hypertension (PA mean pressure at rest >20 mm Hg)
* severe osteoporosis
* severe airway obstruction (FEV1 <50% predicted, FEV1 <60% predicted following bronchodilatation)
* maximum work rate of less than 50 watt during ergometer testing
* uncontrolled asthma
* COPD exacerbation
* severe adipositas (BMI >35 kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 1996-04; Primary Completion 1998-01 (Actual); Study Completion 1998-03 (Actual)

PRIMARY OUTCOMES:
Maximum oxygen uptake | One year
  Maximum oxygen uptake measured during unsteady state cycle ergometer test with work increments of 10 watts each minute until exhaustion.

SECONDARY OUTCOMES:
General quality of life | One year
  Assessment of general quality of life using the german version of the SF-36 questionaire.
Disease-specific quality of life | One year
  Assessment of the disease-specific quality of life using the Asthma Quality of Life Questionnaire (AQLQ)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meyer, M.D., Principal Investigator — Kliniken Mariahilf GmbH, Mönchengladbach, Germany
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Meyer A, Gunther S, Volmer T, Taube K, Baumann HJ. A 12-month, moderate-intensity exercise training program improves fitness and quality of life in adults with asthma: a controlled trial. BMC Pulm Med. 2015 May 7;15:56. doi: 10.1186/s12890-015-0053-8. PMID 25947010